CLINICAL TRIAL: NCT01539668
Title: CareHPV - Hybrid Capture Test on Mobile Unit Program to Improve Cervical Cancer Screening in Brazilian Rural and Remote Areas
Brief Title: Hybrid Capture Test on Mobile Unit Program to Improve Cervical Cancer Screening in Brazilian Rural and Remote Areas
Acronym: careHPV
Status: Completed | Type: Observational
Sponsor: Barretos Cancer Hospital (Other)
Collaborators: QIAGEN Gaithersburg, Inc (Industry)
Responsible Party: Principal Investigator, Adhemar Longatto-Filho, Coordinator, Barretos Cancer Hospital
Other Study IDs: careHPV_2012
Record Dates: First submitted 2012-01-23; First posted 2012-02-27 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-02

CONDITIONS: Cervical Cancer Squamous Cell; Human Papilloma Virus Infection; Human Papilloma Virus-Related Carcinoma; Prevention
Keywords: Cervical Cancer; HPV; Secondary prevention
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cervical cell samples (cytology)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pap sampling: Women who have undergone Pap sampling and HPV and cytology analysis. The samples will be collected in Mobile Units and Non-Mobile Units.

SUMMARY:
This study evaluates the women cervical samples through molecular tests in order to:

1. Deploy the test careHPV (hybrid capture test) in mobile unities of the Barretos Cancer Hospital to evaluate their performance;

DETAILED DESCRIPTION:
Step1: Ambulatory samples First of all the careHPV cervical sample will be collected in specifically tubes, after this, make the cervical sample SurePath collect. Each patient will have two cervical samples. In this moment will be collected 2,000 samples at the Gynecology Department of Barretos Cancer Hospital and the women who be attended in the mobile unit of Barretos surrounding.

Sample1: careHPV The collect will be randomized where 1000 will be collected by the doctor and 1000 by self-sampling. The patient will be oriented by nurse with illustrative material. The self-sampling will be realized like the manufacturing protocol (Qiagen Inc., Gaithersburg, MD).

The cervical sample to cytology (SurePath) will be realized by doctor like a complementary test.

The conditions to store the samples are 15˚C to 30˚C by 2 weeks; 2˚C to 8˚C by 4 weeks; or -20˚C by 2 months to research.

Sample2: SurePath® cytology The cervical sample will be realized like the manufacturing protocol, by doctor. The lamina will be prepared like the equipment manufactory (Becton, Dickinson and Company). The cytological findings will be classifieds like the Bethesda system.

The positives women in careHPV/cytology and the negative careHPV but positive cytology (ASC-US+) will be referred to do the colposcopy (or biopsy) at the Barretos Cancer Hospital.

Step2: Mobiles Unities Samples This step will be collected 3,000 samples to careHPV test and SurePath cytology like a complementary test. The self-sampling won't be made in this step.

The samples will be analyzed in the own mobile unit, during the cities visited. The units involved in the project are that attended Mato Grosso, Goiás, Minas Gerais and Rondônia states, because the significantly number of population assisted.

Step3: HPV genotyping All the positives cases to careHPV test will be submitted to identify the HPV types, then realized at the Molecular Oncology Research Center in the Barretos Cancer Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Any women who come to do the Papanicolaou test at the Barretos Cancer Hospital and in the mobile units on the remote Brazilian areas.

Exclusion Criteria:

* not applicable.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have undegone Pap sampling in a Mobile Unit and Non-Mobile Units.
Sampling Method: Non-Probability Sample
Enrollment: 5079 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
HR-HPV presence in the studied population. | Up to 24 months

SECONDARY OUTCOMES:
The meaning of HPV presence relating with the conventional screening test (Papanicolaou smear), and the pattern of setting cervical lesion (biopsy). | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Adriana T Lorenzi, MSc, Principal Investigator; Adhemar Longatto-Filho, PhD, Study Director — Barretos Cancer Hospital
Locations (1):
- Barretos Cancer Hospital, Barretos, São Paulo, Brazil